CLINICAL TRIAL: NCT03101163
Title: Multicenter, Randomized, Open-Label, Standard Treatment-Controlled Parallel Group Phase 2 Study to Evaluate Efficacy and Safety of Intra-Articular Injections of Autologous Peripheral Blood Stem Cells and Hyaluronic Acid Adjuvant Therapy Following Subchondral Drilling Surgery for the Treatment of Articular Cartilage Injury in the Knee With an Optional Open-Label Extension for the Standard Treatment-Controlled Group
Brief Title: Efficacy and Safety Study of Intra-Articular Injections of Autologous Peripheral Blood Stem Cells Following Subchondral Drilling Surgery for the Treatment of Articular Cartilage Injury in the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KLSMC Stem Cells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLSMC-003
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-03

CONDITIONS: Articular Cartilage Disorder of Knee; Articular Cartilage; Degeneration
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects randomized to the intervention group will undergo subchondral drilling surgery according to standard protocol, and will also receive a regimen of PBSC and HA intra-articular injections and postoperative physiotherapy.
  Interventions: Biological: Autologous peripheral blood stem cells and hyaluronic acid
- Standard treatment (Active Comparator): Subjects randomized to the standard treatment-controlled parallel group will receive intra-articular HA injections and a physiotherapy regimen.
  Interventions: Other: Hyaluronic acid

INTERVENTIONS:
Biological: Autologous peripheral blood stem cells and hyaluronic acid — Regimen of intra-articular PBSC and HA injections and postoperative physiotherapy
  Arms: Intervention
Other: Hyaluronic acid — Regimen of intra-articular HA injections and postoperative physiotherapy
  Arms: Standard treatment

SUMMARY:
This is a 24-month, multicenter, randomized, open-label, standard treatment-controlled, parallel-group, Phase 2 study for adults with large or complicated knee articular cartilage lesions and are candidates for knee joint cartilage repair surgery. The safety and efficacy of intra-articular injections of peripheral blood stem cells (PBSCs) together with hyaluronic acid (HA) after subchondral drilling surgery will be evaluated to determine whether PBSC therapy can improve functional outcome and reduce pain of the knee joint better than a standard treatment (HA injections and physiotherapy regimen).

DETAILED DESCRIPTION:
This is a 24-month, multicenter, randomized, open-label, standard treatment-controlled, parallel-group, Phase 2 study for adults with large or complicated knee articular cartilage lesions and are candidates for knee joint cartilage repair surgery. The safety and efficacy of intra-articular injections of peripheral blood stem cells (PBSCs) together with hyaluronic acid (HA) after subchondral drilling surgery will be evaluated to determine whether PBSC therapy can improve functional outcome and reduce pain of the knee joint better than a standard treatment (HA injections and physiotherapy regimen).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 55 years at screening (20 to 57 years for the open-label extension)
* Present for evaluation and treatment of knee pain, knee swelling, or knee mechanical symptoms due to cartilage lesions
* Provide written informed consent
* International Cartilage Repair Society (ICRS) Grade 3 or 4 lesions diagnosis from MRI scans of the target knee
* All subjects must also satisfy at least 1 of the following inclusion criteria:

  * Isolated knee articular cartilage lesion (single lesion) estimated to be ≥3 cm2 as demonstrated on MRI scanning. Multiple knee articular cartilage lesions (multiple lesions) with at least 1 lesion estimated to be ≥3 cm2 as demonstrated on MRI scanning. Bipolar cartilage defects demonstrated on MRI scanning with at least 1 articular surface lesion to be ≥3 cm2. One or more cartilage defects involving the patello-femoral joint as demonstrated on MRI scanning with at least 1 lesion ≥3 cm2. One or more cartilage defects involving the tibio-femoral joint as demonstrated on MRI scanning with at least 1 lesion to be ≥3 cm2. Previously failed cartilage repair procedures (i.e., microfracture, osteochondral autograft transplantation surgery (OATS), ACI)

Exclusion Criteria:

* Three or more previous surgical interventions on the knee in question.
* Preoperative flexion deformity greater than 10 degrees.
* Presence of ligamentous injury which would require reconstruction, varus or valgus deformity requiring osteotomy, or cases that require complex surgery prior to cartilage regeneration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | 24 months
  Subjective IKDC core as a measure of joint function
Knee injury and Osteoarthritis Outcome (KOOS) pain subdomain | 24 months
  KOOS pain subdomain score as a measure of joint pain

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) for pain | 24 months
  Numeric Rating Scale (NRS) for pain

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Andrews Research & Education Foundation (AREF), Gulf Breeze, Florida, United States
- Kuala Lumpur Sports Medicine Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided